CLINICAL TRIAL: NCT06001073
Title: Prognosis Prediction System of Patients With Cardiovascular and Cerebrovascular Diseases Based on Multi-omics (PROSPECT): a National, Multicenter, Retrospective-prospective, Cohort Study
Brief Title: Prognosis Prediction System of Patients With Cardiovascular and Cerebrovascular Diseases Based on Multi-omics
Acronym: PROSPECT
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Xi'an Gaoxin Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); General Hospital of Ningxia Medical University (Other); Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-353
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease; Arrhythmias, Cardiac; Heart Valve Diseases; Aortic Dissection; Heart Neoplasms; Myocarditis; Hypertension; Cardiomyopathies; Structural Heart Disease; Ischemic Cerebrovascular Disease; Hemorrhagic Cerebrovascular Disease; Brain Neoplasms
Keywords: Cardiovascular diseases; Cerebrovascular diseases; Prognosis; Multi-omics
MeSH Terms: conditions — Coronary Artery Disease; Arrhythmias, Cardiac; Heart Valve Diseases; Aortic Dissection; Heart Neoplasms; Myocarditis; Hypertension; Cardiomyopathies; Brain Neoplasms; Cardiovascular Diseases; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood, feces urine and tissues.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- Coronary artery disease group: Diagnosis of coronary artery disease by clinical guidelines.
  Interventions: Other: Observational; No Interventions were given.
- Arrhythmia group: Diagnosis of arrhythmia by clinical guidelines. by clinical guidelines.
  Interventions: Other: Observational; No Interventions were given.
- Heart valve disease group: Diagnosis of heart valve disease by clinical guidelines.
  Interventions: Other: Observational; No Interventions were given.
- aortic dissection group: Diagnosis of aortic dissection by clinical guidelines.
  Interventions: Other: Observational; No Interventions were given.
- Cardiac masses group: Diagnosis of cardiac messes by clinical guidelines.
  Interventions: Other: Observational; No Interventions were given.
- Myocarditis group: Diagnosis of myocarditis by clinical guidelines.
  Interventions: Other: Observational; No Interventions were given.
- Hypertension group: Diagnosis of hypertension by clinical guidelines.
  Interventions: Other: Observational; No Interventions were given.
- Cardiomyopathy group: Diagnosis of cardiomyopathy by clinical guidelines.
  Interventions: Other: Observational; No Interventions were given.
- Structural heart disease group: Diagnosis of structural heart disease by clinical guidelines.
  Interventions: Other: Observational; No Interventions were given.
- Ischemic cerebrovascular disease group: Diagnosis of ischemic cerebrovascular disease by clinical guidelines.
  Interventions: Other: Observational; No Interventions were given.
- Hemorrhagic cerebrovascular disease group: Diagnosis of hemorrhagic cerebrovascular disease by clinical guidelines.
  Interventions: Other: Observational; No Interventions were given.
- Intracranial space occupying lesion group: Diagnosis of intracranial space occupying by clinical guidelines.
  Interventions: Other: Observational; No Interventions were given.

INTERVENTIONS:
Other: Observational; No Interventions were given. — Observational; No Interventions were given.

SUMMARY:
The etiology and specific pathogenesis of many cardiovascular diseases such as coronary atherosclerosis, cardiomyopathy, atrial fibrillation, and stroke are still unclear. Improving diagnosis and treatment, clarifying the pathogenesis, and providing scientific basis for the prevention and treatment are hot research topics in the study of cardiovascular and cerebrovascular diseases. This study intends to collect clinical data and biological specimen data of patients with cardiovascular and cerebrovascular diseases who meet the inclusion and exclusion criteria, and use multi-omics technology to deeply understand the pathogenic mechanisms of cardiovascular and cerebrovascular diseases and provide new ideas for specific and individualized treatment of patients with cardiovascular and cerebrovascular diseases, to construct early predictive prognostic models and provide a basis for effective treatment of clinical practice in patients with cardiovascular and cerebrovascular diseases.

DETAILED DESCRIPTION:
Cardiovascular and cerebrovascular diseases refer to ischemic and hemorrhagic diseases of the heart, brain and body tissues caused by hyperlipidemia, blood viscosity, atherosclerosis, hypertension, etc. It is one of the major public health problems in the world. The etiology and specific pathogenesis of many cardiovascular diseases such as coronary atherosclerosis, cardiomyopathy, atrial fibrillation, and stroke are still unclear. Improving diagnosis and treatment, clarifying the pathogenesis, and providing scientific basis for the prevention and treatment are hot research topics in the study of cardiovascular and cerebrovascular diseases. This study intends to collect clinical data and biological specimen data of patients with cardiovascular and cerebrovascular diseases who meet the inclusion and exclusion criteria, and use multi-omics technology to deeply understand the pathogenic mechanisms of cardiovascular and cerebrovascular diseases and provide new ideas for specific and individualized treatment of patients with cardiovascular and cerebrovascular diseases, to construct early predictive prognostic models and provide a basis for effective treatment of clinical practice in patients with cardiovascular and cerebrovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are regularly visited and followed up in the appropriate patient; department.
* All patients met at least one of the following diagnostic criteria for cardiovascular and cerebrovascular diseases:
* coronary artery disease group;
* arrhythmia group;
* heart valve disease group;
* aortic dissection group;
* cardiac masses group;
* myocarditis group;
* hypertension group;
* cardiomyopathy group;
* structural heart disease group;
* ischemic cerebrovascular disease group;
* hemorrhagic cerebrovascular disease group;
* intracranial space occupying lesion group.

Exclusion Criteria:

* Age <3 years or >80 years old;
* Pregnant and lactating women;
* The patient declined to provide informed consent to participate in the study;
* None of the above was met, but the patient was temporarily unable to sign the informed consent form due to coma and other reasons, and no legal representative signed it instead. Depending on the patient's condition, the patient may not be able to regain consciousness and sign the informed consent form.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cardiovascular and cerebrovascular diseases will be recruited, including coronary artery disease, arrhythmia, heart valve disease, aortic dissection, cardiac masses, myocarditis, hypertension, cardiomyopathy, structural heart disease, ischemic cerebrovascular disease, hemorrhagic cerebrovascular disease, and intracranial space occupying lesion.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of MACCE | Through study completion, up to 5 years.
  Major adverse cardiovascular and cerebrovascular events, a composite of all-cause mortality, myocardial infarction, coronary revascularization, and stroke.

SECONDARY OUTCOMES:
Change of all-cause mortality | Through study completion, up to 5 years.
  Incidence of patients' death from any cause.
Incidence of myocardial infarction | Through study completion, up to 5 years.
  Changes of serum myocardial zymogram level and ECG were used for diagnosing of myocardial infarction.
Incidence of coronary revascularization. | Through study completion, up to 5 years.
  Incidence of percutaneous coronary intervention or coronary artery bypass grafting.
Incidence of stroke | Through study completion, up to 5 years.
  Stroke were assessed by radiologist using CT scan or other imaging test.

CONTACTS AND LOCATIONS:
Overall Officials: Gouliang Li, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Yang Yan, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiantong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No